CLINICAL TRIAL: NCT03977038
Title: Investigation of Effects of Repetitive Transcranial Magnetic Stimulation (rTMS) on "Hot" and "Cold" Cognitive Systems In Treatment Resistant Depression (TRD)
Brief Title: Investigation of the Effects of Repetitive Transcranial Magnetic Stimulation on Cognition in Depression
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Peter Giacobbe, Clinical Head, Harquail Centre for Neuromodulation, Sunnybrook Health Sciences Centre
Other Study IDs: 096-2019
Record Dates: First submitted 2019-05-23; First posted 2019-06-06 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Major Depressive Disorder; Treatment Resistant Depression
Keywords: Repetitive Transcranial Magnetic Stimulation; Hot Cognition; Cold Cognition; Attentional Imaging; Eye tracking; Cognitive impairment; Cognition
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Cognitive Dysfunction | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — Whole blood specimen will be retained from all participants at 4 time points in the study (Week 0 (baseline), Week 2, Week 6 (last visit) and Week 10 (follow-up)). Bloodwork is obtained in order to monitor for genotype of serotonin transporter polymorphism (5-HTTLPR) , BDNF and potential alterations in the present levels of inflammatory markers of TNF-⍺ and IL-6 involved in the pathophysiological inflammation profile of depression.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- TRD sample: Individuals in the treatment resistant depression (TRD) sample suffer from the condition called TRD. The intervention that will be administered to this group is the standardized rTMS treatment using High Frequency dTMS (HF-dTMS) stimulation over L-DLPFC, at the frequency of 18Hz, at 120% value of the individual's motor threshold, in 5 daily sessions per week, taking place each weekday, over the course of 6 weeks.
  Interventions: Device: repetitive transcranial magnetic stimulation
- Healthy Controls (HC) sample: Individuals in the HC sample are age-, sex-, education-matched to the individuals in the TRD sample. HC sample does not receive any therapeutic treatment and are solely examined as a comparative measure of normal cognitive capabilities.

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — Repetitive transcranial magnetic stimulation (rTMS) is prescribed as first-line treatment for TRD patients (4). rTMS is safe, tolerable and non-invasive neurostimulation procedure where powerful magnetic pulses are transmitted through the skull into the underlying cortical cortex with the aim of electrical current induction within the neural tissue. This study administers a standard dose of rTMS treatment to the TRD patient sample consisting of high frequency deep TMS (HF-dTMS) stimulation over left dorsolateral prefrontal cortex (L-DLPFC), at the frequency of 18Hz, at 120% value of the individual's motor threshold, in 5 daily sessions per week, taking place each weekday, over the course of 6 weeks. The technology of dTMS, which will be used in this study, is an adaptation of the therapeutic intervention of rTMS with the advancement of possessing higher efficacy in targeting deeper brain regions of interest.
  Groups: TRD sample

SUMMARY:
According to the World Health Organization, MDD is attributed as the leading cause of disability worldwide, leaving 300 million individuals affected. Despite the efficacy of pharmacotherapy, a subset of MDD patients, classified as TRD, exhibit suboptimal response and thus require alternative treatment options such as rTMS. Emotional-laden "hot"and Neutral "cold" cognitions are shown to be dysfunctional in depression. Potential pro-cognitive effects remain inconclusive. In this study the investigators seek to investigate whether visual scanning patterns of emotionally laden images may be a biological marker and predictor of rTMS antidepressant efficacy. If so, then changes in visual scanning patterns are expected to precede clinical symptom improvement. Furthermore, changes in visual scanning patterns (which characterizes the state of hot cognition) are compared simultaneously to changes in cold cognition in order to elucidate the neural mechanisms underlying rTMS-induced changes in cognition. It is hypothesized that participants who are responders to rTMS will exhibit a decrease in the amount of time spent looking at dysphoric images will precede clinically detectable changes in mood as measured by a reduction in the scores on the 17-item Hamilton Depression Rating Scale (HDRS-17). The hypothesis for this study corresponds to the alleviation of the dysfunction within the hot cognitive system as a result of rTMS and a potential compensatory effect of cold cognition as a natural reaction of resetting the allocation of cognitive resources.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is prescribed as first-line treatment for patients with Major Depressive Disorder. rTMS is safe, tolerable and non-invasive neurostimulation procedure. rTMS is characterized by an advantage in comparison to traditional pharmacotherapy in the sense that it exerts higher spatial precision in anatomical targeting of the specifically intended brain region compared to medications. The brain region of interest targeted with deep TMS in this study is the left-dorsolateral prefrontal cortex (L-DLPFC) which has been implicated in pathophysiology of depression.

Emotionally-laden functions within the brain are classified as "hot cognition" and contrastingly, affective-neutral areas regulating domains such as concentration, attention, learning and memory and executive function correspond to the characterization of "cold cognition" system. Both ''hot'' (emotion-laden) and ''cold'' (emotion-independent) cognition are known to take a role in the pathophysiology of MDD.

It is known that individuals suffering from depression experience impairments in hot cognition and as a result dedicate excessive focus to negative information, thereby producing negativity bias. A dysfunctional cold cognition system in depression also persists due to hypoactivity and abnormal functional connectivity of its underlying networks. The potential effects of rTMS on hot and cold cognition are currently uncertain. This study seeks to simultaneously evaluate hot and cold cognitive processes in response to deep TMS in order to elucidate the underlying cognitive mechanisms involved. More specifically, the investigators seek to explore the interaction between the two in terms of the time course and magnitude of the improvements in each system in response to TMS, and their relationship to mood improvement.

Methodology The subjects in the TRD group will undergo High Frequency deep TMS (HF-dTMS) stimulation over L-DLPFC, at the frequency of 18Hz, at 120% motor threshold value, for 5 daily sessions per week, over the course of 6 weeks. After the completion of treatment course at the conclusion of the 6 week mark, one post-treatment follow-up visit will take place at 1 month in order to assess any longer-term effects on cognition and depressive symptoms.

* Visual scanning The visual scanning test will consist of the presentation of 81 slides: 32 test slides (consisting of emotional images taken from Karolinska Directed Emotional Faces (KDEF) standardized library of facial expressions as well as a set of images with suicidal valence) and 49 filler slides. Each of the test and filler slides will contain four images at each of the four quadrants of the slide. The subjects' visual scanning behavior of the test slides will be analyzed while the scanning behavior of the filler slides will not be analyzed. Filler slides will change from session to session while the images on the test slides will remain the same. The position as well as the order of presentation of the four images on each test slide will randomly change between sessions. By using a large number of filler slides (different filler slides for each session), a randomized order for the presentation of the test slides and a randomized order for the position of the four images on each test slide, the investigators are aiming to minimize the possibility that patients' scanning behavior will be affected by recall from previous presentations. Each slide will be presented for 11 seconds for a total presentation time of 15 minutes.
* CANTAB measures For measuring the domains of cold cognition, the CANTAB measure which is a series of cognitive tests will be utilized. This battery is comprised of tests in the following cognitive domains: Attention, Executive Function, Memory and Social-Emotional Cognition. For the purposes of this study, the following cognitive tests will be implemented: For the domain of Attention, Motor screening task (MOT) [2 minutes] which evaluates potential sensorimotor or comprehension deficits, and Rapid Visual Information Processing (RVP) [7 minutes] which measures sustained attention are administered. For the domain of Executive Function, One Touch Stockings of Cambridge (OTS) [10 minutes] test that is built upon the foundation of "Tower of Hanoi" test and evaluates working memory and spatial planning subdomains of executive function will be implemented. For the domain of Memory, Verbal Recognition Memory (VRM) [10 minutes] will be used. VRM is a measure of new learning and verbal memory through the ability of collecting verbal information and its retrieval. For the domain of Social-Emotional Cognition, Emotion Recognition Task (ERT) [6-10 minutes] will be utilized which assesses the subject's ability in identification of six basic human emotions in facial expression along that expression's magnitude spectrum. Overall time allocated to conducting the aforementioned CANTAB measures will be approximately 40 minutes. As the subjects are engaging with these tests, the eye-tracking apparatus will be set up in the meantime [15-20 minutes] to enhance efficiency in time management and optimize the use of time. Following the completion of CANTAB tests, the subjects will promptly begin and complete the visual eye-tracking exercise [15 minutes]. Total time allocated to these measures of hot and cold cognition will approximate 1 hour.
* Bloodwork Past research indicates elevated levels of plasma inflammatory markers in depressive patients compared to non-depressed individuals among which markers such as tumor necrosis factor ⍺ (TNF-⍺) and interleukin-6 (IL-6) have been most reliably seen to exhibit heightened concentration levels in plasma. It has also been shown that depressed individuals had a higher likelihood of portraying non-response towards antidepressant medication carry a higher level of inflammatory markers at baseline and follow-up than those who responded to antidepressant therapy.

It has also been suggested that the number of unsuccessful antidepressant treatment trials indicating resistance and non-responsiveness in treatment resistant depressed individuals is associated with elevated plasma concentration of inflammatory markers of TNF-⍺ and IL-6 compared to responsive depressed individuals who had undergone one adequate antidepressant trial successfully and those with no previous history of antidepressant treatment. As a biological marker of rTMS antidepressant efficacy, bloodwork will be obtained a total of 4 times throughout the course of the study in order to monitor for genotype of serotonin transporter polymorphism (5-HTTLPR), brain-derived neurotrophic factor (BDNF) and potential alterations in present levels of the inflammatory markers of TNF-⍺ and IL-6 involved in the pathophysiological inflammation profile of depression.

● Psychiatric scales The severity of depressive symptoms in subjects will be assessed using the physician-rated HDRS-17 and self-report QIDS-SR16 psychiatric scales.

Analysis Following the end of the last visit at Week 6, patients will be grouped by response status: responder, and non-responder. Responder is defined as a patient with a change of 50% or greater on the HDRS-17 measure from baseline (V2) to the last visit (V8).

For each stage of testing, following the start of treatment (i.e. V2 to V8), differences from baseline (V2) of average visual fixation time, average fixation frequency, HDRS-17 and QIDS-SR16 scores will be calculated. The primary outcome measure, i.e., the difference from baseline of the average fixation time measured on different visits (V2 to V8), will be analyzed using linear mixed effect model with fixed effects and a random subject effect. The investigators will initially fit a mixed model with fixed effects of time and group and their interaction, and random intercepts and slopes. Similar models will be built for the secondary outcome variables comprising of average difference from baseline of fixation frequency, HDRS-17 and QIDS-SR16 scores.

The investigators will use the group main effect and the group-time interaction to test the hypothesis that changes in differences from baseline of fixation time differ between responders and non-responders. The investigators expect the differences from baseline of average fixation time will become more negative (decrease) in the responder group but will remain unchanged in the non-responder group. It is also expected that this reduction in the differences from baseline of average fixation time will precede any significant changes in depressive symptom scores on measures of HDRS-17 or QIDS-SR16.

Similarly, changes in the secondary outcome measures (difference from baseline of average fixation frequency, HDRS-17 and QIDS-SR16 scores) during the study course will also be analyzed in order to demonstrate an expected difference between responders and non-responders. The investigators expect the difference from baseline of fixation frequency will increase and that HDRS-17 and QIDS-SR16 will reduce by the conclusion of this study in the responder but not in the non-responder group. The investigators predict, however that any change in the HDRS-17 or QIDS-SR16 scores will succeed visual scanning parameters (i.e., difference from baseline of average fixation time or average fixation frequency) and only be observed at later time points.

ELIGIBILITY:
Inclusion Criteria:

* For the patient group, subjects are required to meet DSM-5 criteria for a diagnosis of Major Depressive Disorder.
* For the healthy control group, subjects should be matched to the patient group in domains of age, sex and education; as well as being devoid of any current or previous history of neuropsychiatric illness.
* Patient group subjects must have a score of at least 20 on the HDRS-17 at time of assessment.
* All subjects (patients and healthy controls) should be between the ages of 18 and 65.
* All subjects (patients and healthy controls) must be capable of providing their informed written consent.
* For the patient group, it is essential that subjects who are taking antidepressant medications maintain a stable dose of medication for at least 4 weeks prior to start of treatment and also continue maintaining this stability throughout the course of treatment.

Exclusion Criteria:

* Subjects suffering from unstable medical conditions
* Subjects with current and past history of epilepsy
* Recent history of substance abuse/dependence (excluding nicotine and caffeine) within the past 6 months as defined by DSM-5
* History of suicide attempts or self-harm within the past 12 months
* Current or previous diagnosis of Bipolar Disorder, Schizophrenia or other psychotic disorders (including psychotic disorder due to general medical condition, substance-induced psychotic, psychotic disorder not otherwise specified) as defined by the MINI
* Previous lack of response to rTMS
* Electroconvulsive therapy (ECT) within the 3 months prior to beginning of study
* Inability to communicate in English language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential TRD participants in this study will be individuals referred by their family doctor or community psychiatrist for diagnostic clarification and/or the provision of treatment options for their mood symptoms. Additionally, individuals who respond to the study advertisement and based on the telephone screening performed by the study physicians, are deemed to meet the study's inclusion and exclusion criteria will be the provision of treatment options for their mood symptoms as well as the opportunity to participate in this study. Healthy Control participants will be age-,sex- and education- matched to the TRD participants and will be representative of the community sample, consisting of healthy individuals with no psychiatric illness.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-05-30 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Change in cold cognition | Participants will be tested once every two weeks for six weeks. To follow up on investigating lasting results, this cognitive battery will be conducted at follow-up at one-month mark (Week 10) from the last visit at Week 6
  Also known as neutral or "non-emotional" cognition, it will be measured by the Cambridge Neuropsychological Test Automated Battery (CANTAB) utilized in the domains of attention, executive function, memory and social/emotional cognition
Change in hot cognition | Participants will be tested once every two weeks for six weeks. To follow up on investigating lasting results, visual stimuli test will be conducted at one-month mark (Week 10) from the last visit at Week 6
  Also known as "emotional" cognition, it will be measured through attentional imaging by an eye tracking task where participants will view image slides presenting images of different valences (emotional, neutral) and the participant's eye gaze estimates will be recorded

SECONDARY OUTCOMES:
depressive symptoms (physician-rated) | TRD participants are assessed for their depressive symptom severity in response to rTMS treatment by the study psychiatrist every two weeks for six weeks, followed by a follow-up visit at one-month mark (Week 10).
  To assess depressive symptom severity in TRD participants, Hamilton Depression Rating Scale (HDRS-17) will be used. HDRS-17 is a 17-item scale, with some items ranging from a score of 0 to 2 points, and some 0 to 4 points. Higher scores represent worse outcome. Total score ranges include: 0-7 considered as "normal", 8-16 categorized as "mild depression", 17-23 as "moderate depression" and above 24 as "severe depression". Minimum score on the scale is 0 and the maximum score on the scale is 52.
depressive symptoms (self-report) | TRD participants are asked to self-report their depressive symptom severity in response to rTMS treatment every two weeks for six weeks, followed by a follow-up visit at one-month mark (Week 10).
  To assess depressive symptom severity in TRD participants, Quick Inventory of Depressive Symptomology (QIDS-SR16) will be used. QIDS-SR16 is a 16-item scale, with each item ranging from score of 0 to 3 points. Higher scores represent worse outcome. Total score ranges include: 0-5 considered as "no depression", 6-10 as "mild depression", 11-15 as "moderate depression", 16-20 categorized as "severe depression" and 21-27 as "very severe depression". Minimum score on the scale is 0 and the maximum score is 27.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Giacobbe, MD, FRCPC, Principal Investigator — Harquail Centre For Neuromodulation, Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Due to confidentiality, IPD will not be shared with other researchers

REFERENCES:
- [Background] Milev RV, Giacobbe P, Kennedy SH, Blumberger DM, Daskalakis ZJ, Downar J, Modirrousta M, Patry S, Vila-Rodriguez F, Lam RW, MacQueen GM, Parikh SV, Ravindran AV; CANMAT Depression Work Group. Canadian Network for Mood and Anxiety Treatments (CANMAT) 2016 Clinical Guidelines for the Management of Adults with Major Depressive Disorder: Section 4. Neurostimulation Treatments. Can J Psychiatry. 2016 Sep;61(9):561-75. doi: 10.1177/0706743716660033. Epub 2016 Aug 2. PMID 27486154
- [Background] World Health Organization. Depression: Fact Sheet. World Health Organization website. http://www.who.int/mediacentre/factsheets/fs369/en/. Updated February 2017.
- [Background] Gupta M, Holshausen K, Best MW, Jokic R, Milev R, Bernard T, Gou L, Bowie CR. Relationships among neurocognition, symptoms, and functioning in treatment-resistant depression. Arch Clin Neuropsychol. 2013 May;28(3):272-81. doi: 10.1093/arclin/act002. Epub 2013 Jan 22. PMID 23343778
- [Background] Roiser JP, Sahakian BJ. Hot and cold cognition in depression. CNS Spectr. 2013 Jun;18(3):139-49. doi: 10.1017/S1092852913000072. Epub 2013 Mar 12. PMID 23481353
- [Background] Rush AJ, Trivedi MH, Wisniewski SR, Nierenberg AA, Stewart JW, Warden D, Niederehe G, Thase ME, Lavori PW, Lebowitz BD, McGrath PJ, Rosenbaum JF, Sackeim HA, Kupfer DJ, Luther J, Fava M. Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR*D report. Am J Psychiatry. 2006 Nov;163(11):1905-17. doi: 10.1176/ajp.2006.163.11.1905. PMID 17074942
- [Background] Harmer CJ, Shelley NC, Cowen PJ, Goodwin GM. Increased positive versus negative affective perception and memory in healthy volunteers following selective serotonin and norepinephrine reuptake inhibition. Am J Psychiatry. 2004 Jul;161(7):1256-63. doi: 10.1176/appi.ajp.161.7.1256. PMID 15229059
- [Background] Stange JP, Jenkins LM, Hamlat EJ, Bessette KL, DelDonno SR, Kling LR, Passarotti AM, Phan KL, Klumpp H, Ryan KA, Langenecker SA. Disrupted engagement of networks supporting hot and cold cognition in remitted major depressive disorder. J Affect Disord. 2018 Feb;227:183-191. doi: 10.1016/j.jad.2017.10.018. Epub 2017 Oct 9. PMID 29100150
- [Background] Robinson OJ, Roiser JP, Sahakian BJ. Hot and cold cognition in depression. In: McIntyre, R.S. (Ed.), Cognitive Impairment in Major Depressive Disorder.Cambridge University Press, Cambridge, UK; 2016.
- [Background] Lantrip C, Gunning FM, Flashman L, Roth RM, Holtzheimer PE. Effects of Transcranial Magnetic Stimulation on the Cognitive Control of Emotion: Potential Antidepressant Mechanisms. J ECT. 2017 Jun;33(2):73-80. doi: 10.1097/YCT.0000000000000386. PMID 28072659
- [Background] Berlim MT, Van den Eynde F, Daskalakis ZJ. High-frequency repetitive transcranial magnetic stimulation accelerates and enhances the clinical response to antidepressants in major depression: a meta-analysis of randomized, double-blind, and sham-controlled trials. J Clin Psychiatry. 2013 Feb;74(2):e122-9. doi: 10.4088/JCP.12r07996. PMID 23473357
- [Background] Serafini G, Pompili M, Belvederi Murri M, Respino M, Ghio L, Girardi P, Fitzgerald PB, Amore M. The effects of repetitive transcranial magnetic stimulation on cognitive performance in treatment-resistant depression. A systematic review. Neuropsychobiology. 2015;71(3):125-39. doi: 10.1159/000381351. Epub 2015 Apr 25. PMID 25925699
- [Background] Cambridge Neuropsychological Test Automated Battery (CANTAB). Cambridge Cognition Ltd Website. https://www.cambridgecognition.com/cantab/
- [Background] Dowlati Y, Herrmann N, Swardfager W, Liu H, Sham L, Reim EK, Lanctot KL. A meta-analysis of cytokines in major depression. Biol Psychiatry. 2010 Mar 1;67(5):446-57. doi: 10.1016/j.biopsych.2009.09.033. Epub 2009 Dec 16. PMID 20015486
- [Background] Howren MB, Lamkin DM, Suls J. Associations of depression with C-reactive protein, IL-1, and IL-6: a meta-analysis. Psychosom Med. 2009 Feb;71(2):171-86. doi: 10.1097/PSY.0b013e3181907c1b. Epub 2009 Feb 2. PMID 19188531
- [Background] Strawbridge R, Arnone D, Danese A, Papadopoulos A, Herane Vives A, Cleare AJ. Inflammation and clinical response to treatment in depression: A meta-analysis. Eur Neuropsychopharmacol. 2015 Oct;25(10):1532-43. doi: 10.1016/j.euroneuro.2015.06.007. Epub 2015 Jun 20. PMID 26169573
- [Background] Haroon E, Daguanno AW, Woolwine BJ, Goldsmith DR, Baer WM, Wommack EC, Felger JC, Miller AH. Antidepressant treatment resistance is associated with increased inflammatory markers in patients with major depressive disorder. Psychoneuroendocrinology. 2018 Sep;95:43-49. doi: 10.1016/j.psyneuen.2018.05.026. Epub 2018 May 19. PMID 29800779
- [Background] Daniele A, Divella R, Paradiso A, Mattioli V, Romito F, Giotta F, Casamassima P, Quaranta M. Serotonin transporter polymorphism in major depressive disorder (MDD), psychiatric disorders, and in MDD in response to stressful life events: causes and treatment with antidepressant. In Vivo. 2011 Nov-Dec;25(6):895-901. PMID 22021682
- [Background] Lee BH, Kim YK. The roles of BDNF in the pathophysiology of major depression and in antidepressant treatment. Psychiatry Investig. 2010 Dec;7(4):231-5. doi: 10.4306/pi.2010.7.4.231. Epub 2010 Nov 23. PMID 21253405
- [Background] Sharp R. The Hamilton Rating Scale for Depression. Occup Med (Lond). 2015 Jun;65(4):340. doi: 10.1093/occmed/kqv043. No abstract available. PMID 25972613
- [Background] Reilly TJ, MacGillivray SA, Reid IC, Cameron IM. Psychometric properties of the 16-item Quick Inventory of Depressive Symptomatology: a systematic review and meta-analysis. J Psychiatr Res. 2015 Jan;60:132-40. doi: 10.1016/j.jpsychires.2014.09.008. Epub 2014 Sep 20. PMID 25300442